CLINICAL TRIAL: NCT00470886
Title: A Non-Interventional, Post-Marketing Surveillance, Phase IV Study to Assess Compliance With Antihypertensive Telmisartan Therapy
Brief Title: Assessment of Compliance With Antihypertensive Telmisartan Therapy
Acronym: COAST
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Bang & Olufsen Medicom (Industry)
Responsible Party: Regional Medical Affairs, Bayer Sp. z o.o.
Other Study IDs: 12827; KL0710PL (Other: Company); 14237 - KL0710SK (Other: Company); NCT00458692 (obsolete NCT alias)
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Telmisartan (Kinzal/Pritor, BAY68-9291)

INTERVENTIONS:
Drug: Telmisartan (Kinzal/Pritor, BAY68-9291) — Primary care clinic hypertensive patients for whom physician decided to start the treatment with telmisartan

SUMMARY:
The purpose of this study is to asses the efficacy and safety of Telmisartan depending on the use of an electronic therapy monitoring device (HelpingHand) in a real life setting and to asses patients compliance to the therapy with Telmisartan in relation to use of electronic therapy monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Untreated or ineffectively treated arterial hypertension

Exclusion Criteria:

* Cholestatic disorders and severe hepatic failure
* Allergy to Telmisartan
* Pregnancy and lactation period
* Unwillingness to participate in the study
* Inability to use the drug reminder device
* Unwillingness to use the drug reminder device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic hypertensive patients for whom physician decided to start the treatment with telmisartan
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of the treatment with telmisartan reported by the physician with regard to usage the HelpingHand device | At all four planned control visits. (Approx. interval between visits 3 months)

SECONDARY OUTCOMES:
Compliance with the treatment calculated on the basis of by HelpingHand and patients questionnaires | At all four planned control visits. (Approx. interval between visits 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Many Locations, Poland
- Many Locations, Slovakia